CLINICAL TRIAL: NCT06333782
Title: Prospective, Multicentric, Single Blind, Randomized Study on the Evaluation of the Safety and Efficacy of Genefill Contour® Versus Comparator in Labia Majora Augmentation
Brief Title: Evaluation of the Safety and Efficacy of Hyaluronic Acid Injection in Labia Majora Augmentation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bioscience Cosmetics SL (Industry)
Collaborators: Eurofins (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-EU-GEN-01; 2023-A02012-43 (Other: ANSM)
Record Dates: First submitted 2023-12-13; First posted 2024-03-27 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Vulvar Atrophy
Keywords: Labia Majora Atrophy; Labia Majora Hypotrophy; Labia Majora Augmentation; Genital rejuvenation

STUDY DESIGN:
Intervention Model Description: Participants would be randomized on two groups: Genefill Contour or comparator (Desirial Plus) at a ratio 1:1
Who Masked: Participant
Masking Description: Single blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Genefill Contour® (Experimental): Participants will be injected with the investigational device Genefill Contour at Visit 1, and Visit 2 only if touch-up needed.
  Interventions: Device: Experimental- Genefill Contour®
- Comparator (Desirial®Plus) (Active Comparator): Participants would be injected with the marketed comparator (Desirial Plus) at Visit 1, and Visit 2 only if touch-up needed.
  Interventions: Device: Marketed comparator - Desirial®Plus

INTERVENTIONS:
Device: Experimental- Genefill Contour® — Genefill Contour® Hyaluronic Acid Injection
  Arms: Genefill Contour®
Device: Marketed comparator - Desirial®Plus — DESIRIAL®PLUS Hyaluronic Acid Injection
  Arms: Comparator (Desirial®Plus)

SUMMARY:
The goal of this interventional clinical investigation using Genefill Contour® CE marked device outside of its indication is to compare with other hyaluronic acid device already marketed for labia majora augmentation in women with labia majora hypotrophy/atrophy.

The primary objective is the evaluation of the safety of Genefill Contour®. The secondary objectives is effectivenes of the investigational device (improvement of patient´s symptoms, patient´s satisfaction, sexual function & pain during injection).

Participants will come to a total of 8 visits (including 2 phone calls) over a period of 12 months. Participants would be enrolled in Genefill Contour® or comparator group.

An ancillary study would be conducted in a cohort of participants evaluating the increase in volume and distance between labia after HA injection

DETAILED DESCRIPTION:
Prospective, Multicentric, Single Blind, Randomized study on the evaluation of the safety and efficacy of Genefill Contour versus comparator in labia majora augmentation. This study analyze the safety and efficacy of the investigational device versus comparator. Participants would be randomized 1:1 between 2 arms (Genefill Contour vs comparator). The study duration is 12 months and will consist in 8 visits (Screening visit, 5 on site visit and 2 phone calls). At week 4, an optional touch-up may be conducted. 110 participants are expected to be included in the trial.

The primary objective is the evaluation of the safety of Genefill Contour®. The secondary objectives is effectivenes of the investigational device (improvement of patient´s symptoms, patient´s satisfaction, sexual function & pain during injection).

An ancillary study would be conducted in a cohort of participants evaluating the increase in volume and distance between labia after HA injection at W4 and W12.

ELIGIBILITY:
Inclusion Criteria:

* Gender: female.
* Age: more than 18 years old.
* Patient affected by labia majora atrophy/hypotrophy as per investigator's judgement and expressing the wish for volume augmentation of the labia majora.
* Patient able to understand and sign the informed consent for study enrolment.
* Patient having given freely and expressly her informed consent.
* Patient affiliated to a health social security system.
* Female of childbearing potential should use a contraceptive regimen recognized as effective since at least 12 weeks before inclusion and during all the study.

Exclusion Criteria:

* Pregnant or breastfeeding woman or planning a pregnancy during the study
* Women who gave birth within 4 months before inclusion.
* Patient who had been deprived of their freedom by administrative or legal decision or who is under guardianship.
* Patient in a social or sanitary establishment.
* Patient suspected to be non-compliant according to the investigator's judgment.
* Patient suffering from a severe or progressive disease.
* Patient with history of auto immune disease.
* Patient immunosuppressed.
* Patient suffering of haemostatic disorder.
* Patient presenting with acute or chronic skin diseases.
* Patient is prone to active inflammatory or infectious processes or presenting clinical signs of inflammation in or close to the labia majora.
* Patient presenting bacterial, fungal or viral infection in or close to labia majora.
* Patient with history of streptococcal disease.
* Patient with recurrent genital herpes (several times a year). A patient asymptomatic in the 6 months before inclusion is eligible.
* Patient with history of pre-cancerous condition or cancer in areas close to the injection site (external urogenital, anal or vaginal).
* Patient with an actual cancer or presence of pre-cancerous cells (vulvar dysplasia).
* Patient with a known tendency to develop keloid or hypertrophic scars.
* Patient with known allergy or hypersensitivity to hyaluronic acid or to one of Genefill Contour, Desirial® Plus, anesthesia (if applicable) and disinfectant components.
* Patient with multiple allergies.
* Patient with a condition or receiving a medication which, in the investigator's judgment, put the patient at undue risk.
* Patient who started oestrogen therapies for treatment of vulvovaginal symptomatology within 3 months before inclusion.
* Patient under treatment for bacterial, fungal or viral infection.
* Patient under treatment with aspirin, anticoagulant, platelets aggregation inhibiting drugs, NSAIDs, immunosuppressive therapy and Vitamin C or treated within one week before inclusion.
* Patient under local hydrating treatment within four weeks before inclusion.
* Patient with history of correction with another resorbable implants with a similar indication within 12 months before inclusion.
* Patient with history of correction with permanent implants including fat graft or semi-permanent in the area of injection.
* Patient who underwent a surgery on labia minora within 12 months before inclusion.
* Patient who underwent a surgery on labia majora at any time.
* Patient having intolerance to gram-positive bacteria.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-05-22 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Mean of number of occurred ADEs (Adverse device effects) | During 4 weeks after injection: from Visit 1 to Visit 2 (week 4) and from Visit 2 (week 4) to week 8 only if Touch-up done at Visit 2.
  Collection of ADEs by patients having received injection with Genefill Contour versus Desirial Plus after 52 weeks of use

SECONDARY OUTCOMES:
Global Aesthetic Improvement Scale (GAIS) assessment by investigator | Week 4, Week 12, Week 24 & Week 52
  Effectiveness of investigational device versus comparator assessed by the investigator using GAIS.
  GAIS score (1-5) as following:
  1 =very much improved 2= Much improved 3=Improved 4= No change 5= Worse
Global Aesthetic Improvement Scale (GAIS) assessment by participant | Week 4, Week 12, Week 24 & Week 52
  Effectiveness of investigational device versus comparator assessed by the participant using GAIS.
  GAIS score (1-5) as following:
  1 =very much improved 2= Much improved 3=Improved 4= No change 5= Worse
Patient (Atrophy/Hypotrophy) symptoms | Week 4, Week 12, Week 24 & Week 52
  Effectiveness of investigational device (Genefill Contour) versus comparator (Desirial Plus) on patient's symptoms.
  A scale from 0 (abscent) to 10 (intolerance) of the following symptoms:
  * Irritation/Burning during daily life
  * Irritation/Burning during sport
  * Iching
  * Stinging
  * Dryness
Sexual function Assessment, The Female Sexual Function Index (FSFI) | Week 4, Week 12, Week 24, Week 36 & Week 52
  Effectiveness of investigational device Genefill Contour) versus comparator (Desirial Plus) on sexual function.
  Patient will be asked about her sexual life, and the answers will be scored from 1 to 5, being 1 as the worst situation and 5 the best.
Patient´s satisfaction | Week 4, Week 12, Week 24, Week 36 & Week 52
  Effectiveness of investigational device (Genefill Contour) versus comparator (Desirial Plus) on patient's satisfaction.
  The patient will be asked about global satisfaction of the treatment and results. The options of the answers are as follows:
  * Very satisfied
  * Satisfied
  * Unsatisfied
  * Very Unsatisfied
Pain during injection-Visual Analogical Scale (VAS) | After the injection at Visit 1 (Day 0) and Visit 2 ( Week 4)
  Pain assessed by participant immediatly after the injection using Visual Analogical Scale (VAS) at Visit 1 and Visit 2 (only if touch-up is needed).
  The rating is from 0 cm (No pain) to 10 cm(Worst pain possible)
Adverse Events collection (Global safety during the study period) | During the whole study, up to 52 weeks
  Collection of unsolicited adverse events from screening Visit to 52 weeks after first injection.
  AE severity range of grades:
  0=mild
  1. moderate
  2. Severe

CONTACTS AND LOCATIONS:
Overall Officials: Dalia Quwaider, PhD, MBA, Study Director — Bioscience Cosmetics
Locations (3):
- France (2):
  - Cabinet renaissance, Levallois-Perret, Paris
  - Palais Flore, Lyon
- Medical Center "Tu sie leczy", Gdansk, Gdansk, Poland

IPD SHARING:
Plan to Share IPD: No